CLINICAL TRIAL: NCT05684159
Title: A Phase II, Open-Label Study of NM8074 in Patients with Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: Study of NM8074 in Patients with AHUS with Evidence of Ongoing Thrombotic Microangiopathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-aHUS-401
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: AHUS - Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Intervention Model Description: The study will enroll a planned total of 12 patients as subjects for the trial, with extra enrollment if needed, at the discretion of the Investigator. All subjects will be assigned to either Cohort 1 or Cohort 2. Enrollment in Cohort 2 will occur after at least three patients in Cohort 1 have been evaluated for safety for 3 days after the first dose. No more than three patients will be dosed in a day. Safety data will be assessed and reviewed by the Sponsor and Study Investigators for dosed subjects prior to dosing of the rest of the study subjects. In Cohort 1, all 6 subjects will be administered 20 mg/kg of NM8074 intravenously every two weeks for a total of 7 doses. All 6 patients in Cohort 2 will receive weekly doses of 10 mg/kg for a total of 4 doses followed by biweekly doses at 20 mg/kg for a total of 5 doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): 6 subjects will receive an intravenous (IV) infusion of NM8074 at every two weeks for a total of 7 doses
  Interventions: Drug: NM8074
- Cohort 2 (Experimental): 6 subjects will receive weekly doses of 10 mg/kg for a total of 4 doses followed by biweekly doses at 20 mg/kg for a total of 5 doses
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. In Cohort 1, all subjects will be administered 20 mg/kg of NM8074 intravenously every two weeks for a total of 7 doses from Day 1 to Day 85 of the Treatment Period. Patients in Cohort 2 will receive weekly doses of 10 mg/kg for a total of 4 doses from Day 1 to Day 22 followed by biweekly doses at 20 mg/kg for a total of 5 doses from Day 29 to Day 85.

SUMMARY:
This is a Phase II, open-label study designed to determine if intravenously administered NM8074 results in remission from TMA in treatment-naïve aHUS patients.

DETAILED DESCRIPTION:
The proposed study, NM8074-aHUS-401,will initially assign six (6) patients per cohort in a 2-cohort trial. In the first cohort, we will evaluate a biweekly dosing regimen whereas in the second cohort, we will evaluate a weekly dose (10 mg/kg) followed by the biweekly dose (20 mg/kg) over a 3-month period. These studies will determine if NM8074 results in remission from TMA in aHUS patients. If the study shows efficacy in aHUS, additional patients may be added per cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years at the time of consent
* Patients with evidence of resistant or relapsed complement-mediated aHUS with symptoms of Thrombocytopenia, hemolysis, ongoing Thrombotic Microangiopathy and acute kidney injury.
* Evidence of ongoing Thrombotic Microangiopathy which includes Haptoglobin <LLN or undetectable and/or presence of schistocytes
* Acute kidney injury (proteinuria/creatinuria > ULN and/or reduced eGFR)
* Platelets less than 150,000 per microliter (Thrombocytopenia)
* Anemia (Hemoglobin ≤10 g/dL) due to hemolysis
* Lactate dehydrogenase (LDH) level ≥ 1.5 times the upper limit of normal (xULN) during Screening
* All patients must be vaccinated prior to dosing with MenACWY Menactra® polysaccharide diphtheria toxoid conjugate vaccination against Neisseria meningitidis serogroups A, C, Y, and W-135 and MenB meningococcal serogroup B vaccine (Bexsero®). If the window of vaccination is short, then patients will be prophylactically treated with appropriate antibiotics
* Willing and able to understand and complete informed consent procedures, including signing and dating the informed consent form (ICF), and comply with the study visit schedule.
* Male patients and partners of child-bearing potential must agree to use contraceptives and male patients must agree to refrain from donating sperm for the duration of the study.
* Female partners of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative pregnancy test at screening and must agree to use highly effective methods of contraception during dosing and for 1 month after stopping the investigational drug.

Exclusion Criteria:

* History of bone marrow, hematopoietic stem cell, or solid organ transplantation
* Treatment with complement blockers
* Patients with infections
* HUS due to ADAMTS-13 deficiency (<5%)
* Kidney disease other than aHUS
* Chronic dialysis (hemo or peritoneal)
* Liver disease or other major autoimmune diseases
* Typical HUS (Shiga toxin +)
* Known Systemic Lupus Erythematosus (SLE), Systemic Sclerosis, or antiphospholipid antibody positivity or syndrome
* History of currently active primary or secondary immunodeficiency
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection within 2 weeks prior to first dose, or history of unexplained, recurrent bacterial infections
* Has a currently active or known history of meningococcal disease or N. meningitidis infection
* Severe concurrent co-morbidities not amenable to active treatment, e.g., patients with severe kidney disease (CKD stage 4, chronic dialysis)
* Females who have a positive pregnancy test result at Screening or on Day 1.
* Pregnant, planning to become pregnant, or nursing female subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Normalization of platelet count (≥150 x 10^9/L) | Up to Study Day 120
Normalization of LDH levels to below ULN | Up to Study Day 120
Normalization of Schistocyte levels (<1%) | Up to Study Day 120
Change from Baseline or Percent Change from Baseline in renal function | Up to Study Day 120
  Assessed via the change from baseline or percent change from baseline in serum creatinine level.
Change from Baseline or Percent Change from Baseline in Haptoglobin | Up to Study Day 120
Change from Baseline or Percent Change from Baseline in Hemoglobin | Up to Study Day 120
Change from Baseline or Percent Change from Baseline in proteinuria/creatininuria | Up to Study Day 120

SECONDARY OUTCOMES:
Time to achieve complete TMA response | Baseline through Study Day 120
Time to achieve higher hemoglobin from baseline | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in blood clots | Up to Study Day 120
Change from Baseline or Percent Change from Baseline in the total number of plasma infusions or exchanges | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in eGFR (estimated glomerular filtration rate) | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in dialysis requirement | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in quality of life (QoL) Assessed via the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale, Version 4. | Baseline through Study Day 120
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale ranging from "Not at all" to "Very much so". All items are summed to create a single fatigue score with a range from 0 to 52 with a better quality of life indicated by a higher score.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Assessed via the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale (QLQ- C30), Version 3.0 | Baseline through Study Day 120
  All EORTC QLQ-C30 scales and single-item measures range from 0 to 100. This includes 3 symptom scales (fatigue, pain, nausea and vomiting), 5 functional scales (physical, role, cognitive, emotional, and social), single-item questions addressing symptoms like insomnia, dyspnea, loss of appetite, and others that are commonly reported by cancer patients, and the perceived financial impact of the disease. A higher score is associated with a greater quality of life for global health status.

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in CP modulation | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in Factor B levels | Baseline through Study Day 120
Change from Baseline or Percent Change from Baseline in plasma concentration of NM8074 | Baseline through Study Day 120
Maximum plasma concentration (Cmax) | Baseline through Study Day 120
Time corresponding to Cmax (tmax) | Baseline through Study Day 120
Area under the drug concentration-time curves (AUC0-t) | Baseline through Study Day 120

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour T, Scully M, Ariceta G, Cataland S, Garlo K, Heyne N, Luque Y, Menne J, Miyakawa Y, Yoon SS, Kavanagh D; 311 Study Group Members. Long-Term Efficacy and Safety of the Long-Acting Complement C5 Inhibitor Ravulizumab for the Treatment of Atypical Hemolytic Uremic Syndrome in Adults. Kidney Int Rep. 2021 Mar 24;6(6):1603-1613. doi: 10.1016/j.ekir.2021.03.884. eCollection 2021 Jun. PMID 34169200
- [Background] Cammett TJ, Garlo K, Millman EE, Rice K, Toste CM, Faas SJ. Exploratory Prognostic Biomarkers of Complement-Mediated Thrombotic Microangiopathy (CM-TMA) in Adults with Atypical Hemolytic Uremic Syndrome (aHUS): Analysis of a Phase III Study of Ravulizumab. Mol Diagn Ther. 2023 Jan;27(1):61-74. doi: 10.1007/s40291-022-00620-3. Epub 2022 Nov 4. PMID 36329366
- [Background] Cofiell R, Kukreja A, Bedard K, Yan Y, Mickle AP, Ogawa M, Bedrosian CL, Faas SJ. Eculizumab reduces complement activation, inflammation, endothelial damage, thrombosis, and renal injury markers in aHUS. Blood. 2015 May 21;125(21):3253-62. doi: 10.1182/blood-2014-09-600411. Epub 2015 Apr 1. PMID 25833956
- [Background] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815